CLINICAL TRIAL: NCT04073108
Title: Causes of Fever of Unknown Origin (FUO) in Infants and Children Attending Assiut University Children Hospital (AUCH)
Brief Title: Causes of FUO in Infants and Children
Status: Unknown | Type: Observational
Last Known Status: Not yet recruiting
Sponsor: Assiut University (Other)
Responsible Party: Principal Investigator, Randa Mohammed Abd El Twab, Principal Investigator, Assiut University
Other Study IDs: cofouoiiacaauch
Record Dates: First submitted 2019-08-03; First posted 2019-08-29 (Actual); Last update posted 2019-08-29 (Actual); Status verified 2019-08

CONDITIONS: Fever of Unknown Origin
MeSH Terms: conditions — Fever of Unknown Origin | interventions — Tuberculin Test

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Diagnostic Test: tuberculin test — tuberclin test used to diagnose tuberculosis as cause of fever of unknown origin

SUMMARY:
Definition: fever < 38˚c for which the cause could not be identified, documented by a health care provider after 3w.evaluation as an outpatient [or after 1w. evaluation in the hospital]. Most cases, however, do not have fever alone, but FUO results from atypical presentation of common diseases. On the other hand FUO lasting longer than 6mo is uncommon in children & suggests granulomatous, autoimmune or auto inflammatory diseases

DETAILED DESCRIPTION:
Fever of unknown origin (FUO) is a relatively common pediatric complaint. The time of FUO generally ranges from 10 to 21 days. Generally the fever should be greater than 38.3 ˚c for at least 10 days with no evident source after initial outpatient or inpatient workup. A broad range of illnesses are known to cause FUO, including infectious, autoimmune and oncologic etiologies. Definitive diagnosis of FUO can be challenging, with many cases resolving spontaneously without a diagnosis. There is currently no standardized diagnostic approach for working up FUO. The general direction of the workup often depends on the patient's presentation, symptoms, and environmental exposures. It is generally accepted that a complete history and physical examination as well as basic laboratory tests, and empiric antibiotic therapy are initial steps in the workup of FUO. With no advanced resources available, radiographs such as chest X-rays and abdominal ultrasonography as well as simple tests e.g. ESR are commonly performed looking for infectious and malignant sources of FUO. If the diagnosis is still obscure laboratory tests for auto immune antibodies or specific infectious agents, are additional logical steps if the diagnosis remains in question.

Unlike adult studies, the categorical distribution of diagnosis of the causes of FUO in pediatrics has not changed in recent decades (Nield&Kamat , 2018) [1]. Additional studies are needed to improve the recognition of causes of prolonged fever in children.

So that FUO is not a single specific medical disorder but may be a potential manifestation of several diseases and disorders. The initial approach to FUO is suggested to be determination of the causes of prolonged fever in each of the body systems, as suggested by the presenting complaint. For instance in the respiratory system in developing countries tuberculosis (TB) must be searched for in the first place. Similarly Protein Energy Malnutrition (PEM), and vitamin D deficiency rickets must be also thought of as a cause of recurrent / chronic chest infection leading to FUO. In the gastrointestinal system persistant/ recurrent diarrhea must be searched for. In the developing countries, urinary tract infection, typhoid fever and viral hepatitis constitute other hidden causes of FUO. Collagen diseases, auto inflammatory diseases as well as immune deficiency diseases and auto immune disorders must be searched for as causes of FUO.

ELIGIBILITY:
Inclusion Criteria:

* All FUO cases admitted to AUCH during one year of the study.

Exclusion Criteria:

* cases of HIV

Ages: 3 Months to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: infants and children
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2019-10-01 (Estimated); Primary Completion 2020-10-01 (Estimated); Study Completion 2021-10-01 (Estimated)

PRIMARY OUTCOMES:
Causes of Fever of unknown origin (FUO) in infants and children attending Assiut University Children Hospital (AUCH) | Baseline
  investigations

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Chien YL, Huang FL, Huang CM, Chen PY. Clinical approach to fever of unknown origin in children. J Microbiol Immunol Infect. 2017 Dec;50(6):893-898. doi: 10.1016/j.jmii.2015.08.007. Epub 2015 Oct 9. PMID 27143687
- [Background] Attard L, Tadolini M, De Rose DU, Cattalini M. Overview of fever of unknown origin in adult and paediatric patients. Clin Exp Rheumatol. 2018 Jan-Feb;36 Suppl 110(1):10-24. Epub 2018 May 3. PMID 29742054
- [Background] Antoon JW, Knudson-Johnson M, Lister WM. Diagnostic approach to fever of unknown origin. Clin Pediatr (Phila). 2012 Nov;51(11):1091-4. doi: 10.1177/0009922811431160. Epub 2011 Dec 12. No abstract available. PMID 22166749
- [Background] Hassan RH, Fouda AE, Kandil SM. Fever of Unknown Origin in Children: A 6 year- Experience in a Tertiary Pediatric Egyptian Hospital. Int J Health Sci (Qassim). 2014 Jan;8(1):13-9. doi: 10.12816/0006067. PMID 24899875